CLINICAL TRIAL: NCT06884436
Title: The Relationship Between Preoperative Cardiology Consultation and the Incidence of Major Adverse Cardiac Events in Patients Without Cardiac Surgery--A Retrospective Cohort Study
Brief Title: Preoperative Cardiology Consultation and the Incidence of Major Adverse Cardiac Events（MACE）
Acronym: MACE
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Jingsheng Lou, Professor, Chinese PLA General Hospital
Other Study IDs: PLAGH-AOC-L05
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Major Adverse Cardiac Events; Acute Myocardial Infarction (AMI); Cardiac Death, Sudden; Cardiac Arrest (CA); Arrhythmia, Cardiac; Heart Failure (HF); Unstable Angina (UA)
Keywords: Cardiology Consultation; Major Adverse Cardiac Events; Preoperative; elderly; electrocardiogram
MeSH Terms: conditions — Cardiovascular Diseases; Death, Sudden, Cardiac; Heart Arrest; Arrhythmias, Cardiac; Heart Failure; Angina, Unstable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Risk Predictors of Major Adverse Cardiac Events: Identify risk factors through the incidence of major adverse cardiac events occurring within 30 days post-surgery, and analyze the benefits to patients through the intervention of cardiology consultations.

SUMMARY:
This cohort study aims to determine when preoperative cardiology consultation is needed to reduce the incidence of major adverse cardiac events (MACE) in elderly patients undergoing non-cardiac surgery. The study collected data on elderly patients with preoperative electrocardiogram (ECG) results who underwent non-cardiac surgery. It was conducted at the First Medical Center of the Chinese People's Liberation Army General Hospital from January 2015 to August 2019. MACE was defined as a composite event occurring within 30 days postoperatively, including acute myocardial infarction, unstable angina, heart failure, new-onset severe arrhythmias, non-fatal cardiac arrest, and cardiac death. Data were extracted using structured query language (SQL) and reviewed by three experienced clinicians. Preoperative cardiology consultation was considered as a mediating variable. By modeling, the confounding factors and risk factors for MACE were identified, and the impact of cardiology consultation as a mediating factor on the incidence of postoperative MACE was evaluated. Additionally, the study aimed to identify which categories of ECG findings necessitate cardiology consultation to reduce the incidence of adverse cardiac events, thereby optimizing the cardiology consultation process.

DETAILED DESCRIPTION:
Background Preoperative electrocardiogram (ECG) is one of the important methods for perioperative assessment. It can reflect the patient's cardiac condition to a certain extent and indicate the potential risk of major adverse cardiac events (MACE). When a patient has an abnormal preoperative ECG, the standard medical procedure is to consult with a cardiologist to assess cardiac risk and adjust cardiac function, thereby reducing the incidence of adverse cardiac events. However, some studies suggest that cardiology consultation may delay surgery for elderly fracture patients and that consultation does not affect the prognosis of some abdominal surgery patients. Conversely, other studies indicate that cardiology consultation can reduce the incidence of adverse cardiac events in patients undergoing major vascular surgery. Additionally, when the patient has a normal ECG, cardiology consultation is usually not provided. Yet, elderly patients often have multiple chronic diseases, and a normal ECG does not completely rule out cardiac problems, which significantly increases the incidence of adverse cardiac events. Therefore, identifying risk factors to reduce the incidence of adverse cardiac events in elderly non-cardiac surgery patients is particularly important.

Objectives:

To investigate the circumstances in which preoperative cardiology consultation is needed to reduce the incidence rate of MACE.

Methods:

MACE was defined as the composite of acute myocardial infarction (MI), unstable angina, heart failure (HF), new-onset severe arrhythmia, nonfatal cardiac arrest, and cardiac death, occurring during or within 30 days following non-cardiac surgery. MACE cases were identified by reviewing medical records. Structured query language (SQL) was employed to extract relevant data elements, including postoperative biochemical tests, electrocardiograms (ECGs), coronary angiograms, postoperative progress notes, and consultation reports. Patients could experience multiple MACE events. Three experienced clinicians conducted independent evaluations of complications. Any discrepancies were resolved through discussion and consensus. This cohort study involved non-cardiac surgery patients from the First Medical Center of the Chinese PLA General Hospital, covering the period from January 2015 to August 2019. Preoperative cardiology consultation was considered as a mediating variable. By modeling, the confounding factors and risk factors for MACE were identified, and the impact of cardiology consultation as a mediating factor on the incidence of postoperative MACE was evaluated. Additionally, the study aimed to identify which categories of ECG findings necessitate cardiology consultation to reduce the incidence of adverse cardiac events, thereby optimizing the cardiology consultation process.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years;
* Preoperative ECG results available.

Exclusion Criteria:

* Age < 65 years;
* Accepted cardiac or neuro surgery;
* Second surgery within 30 days post-operation;
* Patient refused to follow up.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Select elderly patients who underwent elective surgery at the First Medical Center of the PLA General Hospital from January 2015 to August 2019. All subjects will sign an informed consent form; patients who cannot sign the informed consent form will be provided with verbal informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 22000 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
MACE | within 30 days post-surgery
  The entire sample was divided into a development cohort and a validation cohort in a 7:3 ratio. Univariate and multivariate logistic regression analyses were conducted to identify risk predictors of MACE and to establish a nomogram with statistically significant predictors. The development cohort was used to construct the MACE prediction model, while the data from the validation cohort were used for validation. Preoperative cardiology consultation was considered as a mediating variable. By modeling, the confounding factors and risk factors for MACE were identified, and the impact of cardiology consultation as a mediating factor on the incidence of postoperative MACE was evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Jingsheng Lou, PhD & MD, Principal Investigator — The First Medical Center, Chinese PLA General Hospital
Locations (1):
- Department of Anesthesiology, The First Medical Center, Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Given the sensitive nature of the questions posed in this study, we assured participants that their raw data would remain confidential. Therefore, the raw numerical data used to extrapolate the graphs/charts are not present within the manuscript and will not be disclosed. These data will be shared upon reasonable request made to the corresponding author.

REFERENCES:
- [Result] Beattie WS, Lalu M, Bocock M, Feng S, Wijeysundera DN, Nagele P, Fleisher LA, Kurz A, Biccard B, Leslie K, Howell S, Landoni G, Grocott H, Lamy A, Richards T, Myles P; StEP COMPAC Group; Patient Comfort; Clinical Indicators; Delirium Postoperative Cognitive Dysfunction Stroke; Cardiovascular; Data Extractors; Respiratory; Inflammation Sepsis; Acute Kidney Injury; Bleeding Complications Patient Blood Management; Healthcare Resource Utilisation; Patient-Centred Outcomes; Organ Failure and Survival; Cancer Surgery. Systematic review and consensus definitions for the Standardized Endpoints in Perioperative Medicine (StEP) initiative: cardiovascular outcomes. Br J Anaesth. 2021 Jan;126(1):56-66. doi: 10.1016/j.bja.2020.09.023. Epub 2020 Oct 20. PMID 33092804
- [Result] Smilowitz NR, Berger JS. Perioperative Cardiovascular Risk Assessment and Management for Noncardiac Surgery: A Review. JAMA. 2020 Jul 21;324(3):279-290. doi: 10.1001/jama.2020.7840. PMID 32692391
- [Result] Hao L, Xu X, Dupre ME, Guo A, Zhang X, Qiu L, Zhao Y, Gu D. Adequate access to healthcare and added life expectancy among older adults in China. BMC Geriatr. 2020 Apr 9;20(1):129. doi: 10.1186/s12877-020-01524-9. PMID 32272883